CLINICAL TRIAL: NCT00211809
Title: A Controlled Trial of Cognitive-Behavioral Therapy as an Adjunct to Serotonin Reuptake Inhibitors in Body Dysmorphic Disorder
Brief Title: CBT as an Adjunct to SRIs in the Treatment of BDD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 00-0211PS*
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Body Dysmorphic Disorder
Keywords: Body Dysmorphic Disorder; SRIs; Cognitive Behavioral Therapy
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Cognitive Behavioral Therapy; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body dysmorphic disorder (Experimental): Participants with body dysmorphic disorder
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Venlafaxine

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — standard psychiatric evaluation
Drug: Venlafaxine — start dose of 37.5 mg/day and increased to a minimum of 150mg/day, generally over the first 4 weeks and then maintained at that dose for 8 weeks.
  Other Names: Effexor

SUMMARY:
The research project is a controlled pilot study of the efficacy of cognitive-behavioral therapy (CBT) as an adjunct to serotonin reuptake inhibitor (SRI) pharmacotherapy in body dysmorphic disorder (BDD). This study assesses the efficacy of CBT in comparison to relaxation and stress management training (RSMT), an active control treatment

DETAILED DESCRIPTION:
In total, 20 BDD patients aged 16 through 65 will participate. To be eligible they must meet DSM-IV criteria for BDD, have a score of 20 or greater on the BDD modification of the Yale Brown Obsessive-Compulsive Scale (BDD-YBOCS) and be on a stable, therapeutic does of an SRI (at least 12 weeks on the SRI with 8 weeks at a therapeutic dose: acceptable medications (therapeutic daily doses) are citalopram (40mg), clomipramine (150mg), fluoxetine (40mg), fluvoxamine (150mg), paroxetine (40mg), sertraline (50mg), and venlafaxine (150mg).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65
* A diagnosis of DSM-IV BDD or its delusional variant (delusional disorder, somatic type)
* Ability to communicate meaningfully with the investigators
* Competent to provide written consent, if over 18 years old, or competent to provide written assent, if 16-17 years, 11 months
* Parental consent, if under 18 years old
* For phase two: must be on a stable therapeutic dose of one of the following SRI medications for at least 8 weeks: fluoxetine, fluvoxamine, venlafaxine, clomipramine, paroxetine, citalopram, or sertraline.

Exclusion Criteria:

* current or lifetime diagnosis of any DSM_IV psychotic disorder not attributable to delusional BDD, current or lifetime diagnosis of DSM-IV bipolar disorder,
* current or recent (within 2 months of study entry) DSM-IV alcohol or substance dependence or abuse,
* recent suicide attempt, or suicidal ideation that warrants consideration of hospitalization,
* need for inpatient or partial hospital treatment,
* use of any medication prescribed for the treatment of BDD other than SRIs, including tricyclic antidepressants, buspirone, or neuroleptics,
* presence of any significant and/or unstable medical condition,
* females who are pregnant or breast-feeding, or who are sexually active and not using adequate contraception.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Andrea Allen, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Allen A, Hadley SJ, Kaplan A, Simeon D, Friedberg J, Priday L, Baker BR, Greenberg JL, Hollander E. An open-label trial of venlafaxine in body dysmorphic disorder. CNS Spectr. 2008 Feb;13(2):138-44. doi: 10.1017/s1092852900016291. PMID 18227745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by advertising and other media and by referral from outside clinicians.
Groups:
- Body Dysmorphic Disorder: Participants with body dysmorphic disorder
  Standard Psychiatric Evaluation
  Venlafaxine: start dose of 37.5 mg/day and increased to a minimum of 150mg/day, generally over the first 4 weeks and then maintained at that dose for 8 weeks.
Period: Overall Study
Arm/Group | Body Dysmorphic Disorder
Started | 17
Completed | 11
Not Completed | 6
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 2
Not completed — Pregnancy | 1
Not completed — side effects | 2

BASELINE CHARACTERISTICS:
Arm/Group | Body Dysmorphic Disorder
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
SSRI history [Count of Participants; unit: Participants]
  SSRI naive | 7
  prior failed SSRI trials | 10

OUTCOME MEASURES:

1. Primary Outcome: Body Dysmorphic Disorder Examination
Description: Body Dysmorphic Disorder Examination - Self Reported (BDDE-SR) score - The BDDE-SR is a 30-item self-rating of BDD symptoms, with a more specific measure of body image dissatisfaction. Each item is rated 0 (no dissatisfaction to 6 (extreme dissatisfaction), with total score from 0 to 180.
Time Frame: baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Participants with Body Dysmorphic Disorder at baseline
- Endpoint: Participants with Body Dysmorphic Disorder after Venlafaxine treatment up to 16 weeks
Arm/Group | Baseline | Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale | 113.91 (27.41) | 107.73 (39.93)

2. Primary Outcome: Yale Brown Obsessive Scale
Description: Yale Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS) - a 12-item semistructured clinician-rated instrument designed to rate severity of body dysmorphic disorder (BDD) symptoms during the past week. The score for each item ranges from 0 (no symptoms) to 4 (extreme symptoms). The BDD-YBOCS Obsession Subtotal score range is 0-20 and the BDD-YBOCS Compulsion Subtotal score range is 0-20. The BDD-YBOCS Insight/Avoidance Subtotal score range is 0-8. The total BDD-YBOCS score range is from 0 (not present or extremely mild) to 48 (severe). Each item is rated as a composite of all the patient's appearance related obsessions and compulsive behaviors independent of their content.
Time Frame: baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale
  Psychiatrist's Ratings for Total | 34.64 (5.09) | 26.55 (11.28)
  Psychiatrist's Ratings for Obsessions | 14.73 (2.20) | 11.45 (5.03)
  Psychiatrist's Ratings for Compulsions | 14.82 (1.20) | 11.55 (4.93)
  Psychologist's Ratings for Total | 35.91 (4.21) | 28.27 (9.49)
  Psychologist's Ratings for Obsessions | 14.45 (4.57) | 12.09 (4.72)
  Psychologist's Ratings for Compulsions | 16.09 (2.30) | 12.18 (3.84)

3. Primary Outcome: Body Dysmorphic Disorder Clinical Global Impressions Scale
Description: The Clinical Global Impression-Improvement Scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Body Dysmorphic Disorder: Participants with body dysmorphic disorder after Venlafaxine treatment up to 16 weeks
Arm/Group | Body Dysmorphic Disorder
Number analyzed (Participants) | 11
units on a scale
  Psychiatrist's Ratings | 2.73 (0.91)
  Psychologist's Ratings | 3.00 (1.00)

4. Secondary Outcome: Brown Assessment of Beliefs Scale
Description: The Brown Assessment of Beliefs Scale (BABS) rates the degree of conviction and insight patients have concerning their beliefs. The BABS consists of 7 items: the first 6 items are added to obtain the total BABS score. An additional item (ideas of reference) is not included in the total score. Scoring is from 0 (least severe) to 4 (most severe), with total score from 0 to 24.
Time Frame: Baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale
  Psychiatrist's Ratings | 15.82 (5.19) | 16.91 (4.70)
  Psychologist's Ratings | 15.91 (6.47) | 14.82 (6.46)

5. Secondary Outcome: Beck Depression Inventory II
Description: The Beck Depression Inventory II (BDI-II) is a 21 item self-report inventory measuring the severity of depression. Individuals are asked to respond to each question based on a two-week time period. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms.
Time Frame: Baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale | 28.77 (11.49) | 22.18 (15.30)

6. Secondary Outcome: Beck Anxiety Inventory
Description: The Beck Anxiety Inventory (BAI) is a 21-question multiple choice, self-report inventory that is used for measuring the severity of anxiety. Scoring is from a 0 (not at all) to 3 (severe) with a total score range of 0-63. Higher total scores indicate more severe anxiety symptoms.
Time Frame: Baseline and up to 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | Endpoint
Number analyzed (Participants) | 11 | 11
units on a scale | 16.90 (8.23) | 12.55 (10.86)

ADVERSE EVENTS:
Arm/Group | Body Dysmorphic Disorder
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
The primary limitations of this study are the small sample size, the open-label design, and the primarily female sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes